CLINICAL TRIAL: NCT06345898
Title: Clinical Study on the Safety and Efficacy of JWK002 Injection Administered as a Single Subretinal Injection in Subjects With X-linked Retinoschisis
Brief Title: Safety and Efficacy of a Single Subretinal Injection of JWK002 Gene Therapy in Subjects With X-linked Retinoschisis(XLRS)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Fang Lu, Professor, West China Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-1479
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: X Linked Retinoschisis
Keywords: X Linked Retinoschisis
MeSH Terms: conditions — Retinoschisis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JWK002 at Low Dose Group (Experimental): Subretinal injection low dose of JWK002 in one eye
  Interventions: Drug: JWK002
- JWK002 at Medium Dose Group (Experimental): Subretinal injection medium dose of JWK002 in one eye
  Interventions: Drug: JWK002

INTERVENTIONS:
Drug: JWK002 — Subretinal administration of gene therapy vector JWK002 to one eye.

SUMMARY:
This trial is to evaluate the safety and efficacy of JWK002 treatment of X-linked retinoschisis(XLRS). This study will enroll subjects aged 5-18 years old to receive a sub-retinal injection of JWK002.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the purpose and requirements of the trial, voluntarily participate in the clinical trial and sign the informed consent, and be able to cooperate with the testing required in various studies according to the requirements of the program;
2. Male, ≥5 years old and < 18 years old (subject to the date of signing the informed consent);
3. Clinically diagnosed XLRS, identified by genetic testing as RS1 gene mutation, and do not carry other mutations causing ophthalmic genetic diseases;
4. Best corrected visual acuity (BCVA) of the study eye ≤63 letters (equivalent to Snellen 20/63); Best corrected visual acuity (BCVA) ≥34 letters (equivalent to Snellen 20/200).

Exclusion Criteria:

1. Carbonic anhydrase inhibitor treatment within 3 months;
2. The presence of other conditions in the study eye that may cause vision loss (e.g., atrophy of the optic nerve, advanced glaucoma, uveitis, the presence of vesicular splitting chambers or vesicular retinal detachment that may affect the subretinal injection operator);
3. Those who study the retinal observation and examination caused by lens, cornea or other refractive interstitial turbidity;
4. There are eye conditions affecting subretinal injection or eye conditions affecting the determination of the study endpoint;
5. Patients who had undergone internal eye surgery within 6 months;
6. Patients with AAV8 neutralizing antibody titer ≥1:1000;
7. Have previously received any gene therapy or cell therapy;
8. fertile subjects are unwilling to use contraception;
9. The presence of any of the following: an active infection that the investigator believes may affect the patient's participation in the study or affect the study results that requires systematic treatment; Hepatitis B surface antigen positive, hepatitis B virus deoxyribonucleic acid (HBV DNA) copy number > ULN; Hepatitis C virus (HCV) antibody positive and HCV-RNA copy number >ULN; Treponema pallidum antibody positive; Positive for human immunodeficiency virus (HIV) antibodies;
10. Malignant tumors (basal cell or squamous cell skin cancer) were diagnosed within 5 years prior to screening;
11. has or has had a systemic immune system disease;
12. Laboratory values considered to be clinically significant were abnormal: alanine and/or aspartate transaminase >2.5×ULN, total bilirubin >1.5×ULN, serum creatinine >1.5×ULN, prothrombin time ≥1.5×ULN, activated partial thromboplastin time ≥1.5×ULN; (13) have a severe allergy or a known allergy to the drugs used in the treatment or examination in the study protocol, including the investigational drug allergy;

(14) Other situations that the investigator considers inappropriate for participation in this study.

Ages: 5 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2033-11-30 (Estimated); Study Completion 2033-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety(Participants With Ocular and Non-ocular AEs (Adverse Events) and SAEs (Serious Adverse Events) | baseline to day 7, day 14, month 1, 3, 6, 12
  The primary outcome measures are safety, determined by the number of ocular and non-ocular Study Drug-related adverse events (SDAE), treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs).

SECONDARY OUTCOMES:
Best corrected visual acuity (BCVA) | baseline to day 7, day 14, month 1, 2, 3, 6, 12
  Visual acuity of the study eye was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS)
Full-field electroretinogram(ff-ERG) | baseline to month 1, 3, 6, 12
  The ERG measurement will be performed based on the standards of international society for clinical electrophysiology of vision (ISCEV).
Macular structure as assessed by swept source optical coherence tomography | baseline to month 1, 3, 6, 12
  Change in swept source optical coherence tomography(SS-OCT)
Visual field | baseline to month 1, 3, 6, 12
  Change in visual field assessed by Humphrey perimetry

CONTACTS AND LOCATIONS:
Overall Officials: Fang Lu, Principal Investigator — lufang@wchscu.cn
Locations (1):
- West China Hospital, Chengdu, Sichuan, China